CLINICAL TRIAL: NCT00085982
Title: Phase II Trial of Effect of Metreleptin Therapy in Severe Insulin Resistance
Brief Title: Effect of Metreleptin Therapy in the Treatment of Severe Insulin Resistance
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 030257; 03-DK-0257
Record Dates: First submitted 2004-06-18; First posted 2004-06-21 (Estimated); Results first posted 2021-12-15 (Actual); Last update posted 2025-01-30 (Actual); Status verified 2024-12

CONDITIONS: Severe Insulin Resistance
Keywords: Rabson Mendenhall; Type B Insulin Resistance; Type A Insulin Resistance
MeSH Terms: conditions — Insulin Resistance; Diabetes Mellitus, Insulin-Resistant, with Acanthosis Nigricans | interventions — metreleptin

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Leptin Treatment (Experimental): 300 mg of study drug administered via subcutaneous (SC) injections.
  Interventions: Drug: Metreleptin

INTERVENTIONS:
Drug: Metreleptin — Administered SC twice/day to achieve physiological concentrations that will be effective in improving the severe state of insulin resistance seen in patients with genetic defects on their insulin receptor mutation

SUMMARY:
Study Description:

Patients with mutations of the insulin receptor have diabetes that is challenging to control with conventional therapies, leading to early morbidity and mortality. We hypothesize that recombinant leptin (metreleptin) in these patients will improve glycemia control.

Objectives:

Primary Objective: To determine if 1 year of metreleptin will improve glycemia control in patients with genetic defects of the insulin receptor. Secondary Objectives: To determine mechanisms by which metreleptin improves glycemia.

Endpoints:

Primary Endpoint: Hemoglobin A1c.

Secondary Endpoints: fasting plasma glucose, fasting insulin/C-peptide, glucose/insulin/C-peptide area under the curve during oral glucose tolerance test.

Study Population:

20 male or female patients with mutations of the insulin receptor, age (Bullet)5 years, at the NIH Clinical Center.

Description of Sites/Facilities Enrolling Participants: Description of Study Intervention:

NIH Clinical Center

Open label study of metreleptin, 0.2 mg/kg/day (max dose 0.24 mg/kg/day).

DETAILED DESCRIPTION:
Study Description:

Patients with mutations of the insulin receptor have diabetes that is challenging to control with conventional therapies, leading to early morbidity and mortality. We hypothesize that recombinant leptin (metreleptin) in these patients will improve glycemia control.

Objectives:

Primary Objective: To determine if 1 year of metreleptin will improve glycemia control in patients with genetic defects of the insulin receptor. Secondary Objectives: To determine mechanisms by which metreleptin improves glycemia.

Endpoints:

Primary Endpoint: Hemoglobin A1c.

Secondary Endpoints: fasting plasma glucose, fasting insulin/C-peptide, glucose/insulin/C-peptide area under the curve during oral glucose tolerance test.

Study Population:

20 male or female patients with mutations of the insulin receptor, age (Bullet)5 years, at the NIH Clinical Center.

Description of Sites/Facilities Enrolling Participants: Description of Study Intervention:

NIH Clinical Center

Open label study of metreleptin, 0.2 mg/kg/day (max dose 0.24 mg/kg/day).

ELIGIBILITY:
* INCLUSION CRITERIA:
* Provision of signed and dated informed consent form
* Male or female, aged > 5 years
* Clinically significant, severe insulin resistance caused by a known or suspected defect in the insulin receptor
* Presence of at least one of the following metabolic abnormalities:

  * Fasting insulin >30 micro U/ml, or
  * Presence of diabetes as defined by the 2006 American Diabetes Association (ADA) criteria:

    * Fasting plasma glucose >= 126 mg/dL
    * 2 hour plasma glucose >= 200 mg/dL following a 75 gram (1.75g/kg if less than 40kg) oral glucose load, or
    * Diabetic symptoms with a random plasma glucose >= 200 mg/dL

EXCLUSION CRITERIA:

* Pregnant at time of enrollment, women in their reproductive years who do not use an effective method of birth control, and women currently nursing or lactating within 6 weeks of having completed nursing.
* Known infectious liver disease
* Known HIV infection
* Current alcohol or substance abuse
* Active tuberculosis
* Use of anorexigenic drugs
* Other conditions which in the opinion of the clinical investigators would impede completion of the study.
* Subjects who have a known hypersensitivity to E. Coli derived proteins.

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2003-08-21 (Actual); Primary Completion 2019-10-23 (Actual); Study Completion 2030-01-01 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca J Brown, M.D., Principal Investigator — National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Sekizkardes H, Chung ST, Chacko S, Haymond MW, Startzell M, Walter M, Walter PJ, Lightbourne M, Brown RJ. Free fatty acid processing diverges in human pathologic insulin resistance conditions. J Clin Invest. 2020 Jul 1;130(7):3592-3602. doi: 10.1172/JCI135431. PMID 32191645
- [Derived] Okawa MC, Tuska RM, Lightbourne M, Abel BS, Walter M, Dai Y, Cochran E, Brown RJ. Insulin Signaling Through the Insulin Receptor Increases Linear Growth Through Effects on Bone and the GH-IGF-1 Axis. J Clin Endocrinol Metab. 2023 Dec 21;109(1):e96-e106. doi: 10.1210/clinem/dgad491. PMID 37595266
- [Derived] Okawa MC, Cochran E, Lightbourne M, Brown RJ. Long-Term Effects of Metreleptin in Rabson-Mendenhall Syndrome on Glycemia, Growth, and Kidney Function. J Clin Endocrinol Metab. 2022 Feb 17;107(3):e1032-e1046. doi: 10.1210/clinem/dgab782. PMID 34718628
- [Derived] Brown RJ, Cochran E, Gorden P. Metreleptin improves blood glucose in patients with insulin receptor mutations. J Clin Endocrinol Metab. 2013 Nov;98(11):E1749-56. doi: 10.1210/jc.2013-2317. Epub 2013 Aug 22. PMID 23969187
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2003-DK-0257.html

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Leptin Treatment
Started | 11
Completed | 5
Not Completed | 6

BASELINE CHARACTERISTICS:
Groups:
- Leptin Treatment: 300 mg of study drug administered via SC injections.
  Metreleptin: Administered SC twice/day to achieve physiological concentrations that will be effective in improving the severe state of insulin resistance seen in patients with genetic defects on their insulin receptor mutation
Arm/Group | Leptin Treatment
Number analyzed (Participants) | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 13.12 (5.47)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 8
  Unknown or Not Reported | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: African | 1
  Race: Asian | 1
  Race: Caucasian | 7
  Race: Filipino | 2
A1c [Mean (Standard Deviation); unit: percent] | 10.38 (1.17)
Fasting blood glucose [Mean (Standard Deviation); unit: mg/dL] | 155.27 (71.22)
Fasting Insulin [Mean (Standard Deviation); unit: mcU/mL] | 597.26 (787.15)

OUTCOME MEASURES:

1. Primary Outcome: Change in HbA1C
Description: Change in HbA1C at month 12 from baseline.
Time Frame: Change at month 12 from baseline
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | Leptin Treatment
Number analyzed (Participants) | 11
percent | -0.336 (1.921)

2. Secondary Outcome: Change in Fasting Insulin Level
Description: Change in fasting insulin level at month 12 from baseline
Time Frame: Change at month 12 from baseline
Measure: Mean (Standard Deviation); unit: mcU/mL
Arm/Group | Leptin Treatment
Number analyzed (Participants) | 11
mcU/mL | -58.31 (85.21)

3. Secondary Outcome: Change in Fasting Blood Glucose
Description: Change in fasting blood glucose at month 12 from baseline.
Time Frame: Change at month 12 from baseline
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Leptin Treatment
Number analyzed (Participants) | 11
mg/dL | -6.91 (86.1)

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Leptin Treatment
All-Cause Mortality (participants affected / at risk) | 0/11
Serious Adverse Events (participants affected / at risk) | 5/11
Other Adverse Events (participants affected / at risk) | 7/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Leptin Treatment (N=11)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
Brain lesion (Nervous system disorders) | 1 (1)
DKA (Endocrine disorders) | 2 (3)
Edema (General disorders) | 1 (1)
Hyperglycemia (Endocrine disorders) | 1 (1)
papillary carcinoma of thyroid (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Seizure (Nervous system disorders) | 1 (1)
Septic shock (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Leptin Treatment (N=11)
Acrochordon (Skin and subcutaneous tissue disorders) | 1 (1)
Alcohol withdrawal (Psychiatric disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1)
Candidiasis (Infections and infestations) | 1 (1)
Cataract (Eye disorders) | 1 (1)
Cerumen impaction (Ear and labyrinth disorders) | 1 (1)
Cholesteatoma (Ear and labyrinth disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
COVID-19 (Infections and infestations) | 1 (1)
Cracked tooth (Musculoskeletal and connective tissue disorders) | 1 (1)
Dental abscess (Infections and infestations) | 2 (2)
Depression (Psychiatric disorders) | 1 (2)
Edema (General disorders) | 1 (1)
Elevated lactate (Metabolism and nutrition disorders) | 1 (1)
GERD (Gastrointestinal disorders) | 1 (1)
Glaucoma (Eye disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 2 (2)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1)
Indigestion (Gastrointestinal disorders) | 1 (1)
Ketosis (Metabolism and nutrition disorders) | 1 (1)
Kidney stone (Renal and urinary disorders) | 1 (2)
Mastoidectomy & tympanostomy tube placement (Surgical and medical procedures) | 1 (1)
Mitral & tricupsid valve regurgitation (Cardiac disorders) | 1 (1)
Pain (General disorders) | 1 (1)
Seizure (Nervous system disorders) | 1 (4)
Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Throid nodule (Endocrine disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Weight loss (Metabolism and nutrition disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-05-05): https://cdn.clinicaltrials.gov/large-docs/82/NCT00085982/Prot_SAP_000.pdf